CLINICAL TRIAL: NCT02590250
Title: Evaluation of the Safety and Effectiveness of BOTOX® (Botulinum Toxin Type A) in the Treatment of Patients With Urinary Incontinence Due to Neurogenic Detrusor Overactivity or Overactive Bladder: A Phase IV Non-interventional Post-marketing Surveillance Study in India
Brief Title: A Safety and Efficacy Study of BOTOX® (Botulinum Toxin Type A) in Patients With Urinary Incontinence Due to Neurogenic Detrusor Overactivity or Overactive Bladder in India
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-140
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BOTOX®: Patients who receive botulinum toxin Type A (BOTOX®) treatment for Neurogenic Detrusor Overactivity or Overactive Bladder as per local standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A treatment for Neurogenic Detrusor Overactivity or Overactive Bladder as per local standard of care in clinical practice.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This is a Post-Marketing Surveillance study in India to evaluate safety and efficacy of BOTOX® (Botulinum Toxin Type A) in the treatment of patients with urinary incontinence due to neurogenic detrusor overactivity or overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urinary incontinence due to NDO or OAB treated with BOTOX® as per local standard of care in clinical practice.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with urinary incontinence (due to NDO, eg, as a result of SCI or MS, or due to OAB) who have an inadequate response to or are intolerant of an anticholinergic medication
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Change from the baseline value of the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | at up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahunna Ukah, Study Director — Allergan
Locations (12):
- India (12):
  - NU Hospitals, Padmanabha Nagar, Banglore
  - Bodyline Hospitals, Ahmedabad, Gujarat
  - Fortis Hospitals, Bengaluru, Karnataka
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute, Mumbai, Maharashtra
  - AMAI Charitable Trust's ACE Hospital and Research Centre, Pune, Maharashtra
  - Inamdar Multispeciality Hospital, Pune, Maharashtra
  - Dr. Ram Manohar Lohia Hospital, New Delhi, National Capital Territory of Delhi
  - Indian Spinal Injuries Centre, New Delhi, National Capital Territory of Delhi
  - Fortis Escorts Heart Institute, Okhla Road, New Delhi
  - Christian Medical College & Hospital, Ludhiana, Punjab
  - Christian Medical College and Hospital, Vellore, Tamil Nadu
  - Global Hospital, Hyderabad, Telangana

REFERENCES:
- See also: More Information — http://AllerganClinicalTrials.com